CLINICAL TRIAL: NCT03472794
Title: Adaptation of a Knowledges Exchange Portal (KEP) Between Healers and Patients : Study of Obstacles and Sources to the Use of a KEP in the Case of Women Affected by a Breast Cancer in Nouvelle Aquitaine(Sav-AQ)
Brief Title: Adaptation of a Knowledges Exchange Portal Between (KEP) Healers and Patients : Obstacles and Sources to KEP Use for Breast Cancer Women
Acronym: Sav-AQ
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: SRIOP 2016, SIRIC BRIO (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/19
Record Dates: First submitted 2018-01-31; First posted 2018-03-21 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: web portal: " Mon réseau cancer du sein " ("My Breast cancer Network") — web portal: " Mon réseau cancer du sein "

SUMMARY:
The project is imbued with the whole problematic of patient follow-up and patient support, taking into account the experiences and needs of breast cancer patients. It concerns the dissemination of knowledge through the implementation of a specific clinical innovation designed to optimizing breast cancer patient pathway. The " Patients en réseau " association offers us to participate at the web platform evolution Mon Réseau Cancer du Sein in adapting it. The feasibility study focuses on (1) the platform utilization and (2) sources and obstacles to its utilization in the French context

DETAILED DESCRIPTION:
One of the French Cancer Plan 2014-2019 objectives is to improve the town-hospital coordination and information's exchange between professionals. This research project aims to reach this important objective of exchange development and the amelioration of the coordination concerning breast cancer women. Breast cancer requires the integration of aggressive treatments implying physical, psychological and social consequences. That's why an optimized care pathway needs a coordinated and multidisciplinary organization, and more particularly a personalized approach taking into account the whole patients' needs in physical, psychological and social perspectives. To reach this goal, it is important to support those patients, to answer their needs for a better disease management in their own health pathways. The research issues lie in this outcome.

The project is imbued with the whole problematic of patient follow-up and patient support, taking into account the experiences and needs of breast cancer patients. It concerns the dissemination of knowledge through the implementation of a specific clinical innovation designed to optimizing breast cancer patient pathway.

The " Patients en réseau " association offers us to participate at the web platform evolution Mon Réseau Cancer du Sein in adapting it. The feasibility study focuses on (1) the platform utilization and (2) sources and obstacles to its utilization in the French context

ELIGIBILITY:
Inclusion criteria of patients :

* Age ≥ 18 y.o;
* With a diagnosis of breast cancer,
* treated at the Bergonié Institute;
* Patients who express a non-opposition to participate to SAVAQ research;
* Patients who have an Internet access at home.

Inclusion criteria of healers :

- Doctors, Nurse, Senior health manager, Technologist medical imaging from the center participated to the research

Exclusion criteria of patients:

* Patients with a severe psychiatric pathology (medical diagnosis);
* Patients who doesn't speak French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 women with a breast cancer will participate to the study, they will represent a sufficient and realis effective considering the active list of treated patients with a breast cancer at the Bergonié Institute.
  5 healers (one nurse, two doctors, a senior health manager, a manipulator in medical imaging)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Feasability of the web portal | Month 6
  Number of connections to the portal each month:
  * Types of documents consulted
  * Types of downloaded documents
  * Types of documents sought
  * Connection duration
  * Number of connections
  * Number of comments / questions posted
  * Number of comments / questions viewed
  * Number of comments / questions sought

SECONDARY OUTCOMES:
Number of the portal connections realized each month | Month 6
  Number of the portal connections realized each month
Number of webpages used | Month 6
  Number of webpages used
Number of status posted | Month 6
  Number of status posted
Number of comments/questions posted | Month 6
  Number of comments/questions posted
Number of "like" emoticon posted | Month 6
  Number of "like" emoticon posted
Number of "comfort" emoticon posted | Month 6
  Number of "comfort" emoticon posted
Number of "favorites" emoticon posted | Month 6
  Number of "favorites" emoticon posted
Number of "mood" posted | Month 6
  Number of "mood" posted
Number of private posts posted | Month 6
  Number of private posts posted
Number of webpages consulted | Month 6
  Number of webpages consulted
Number of leaflets consulted | Month 6
  Number of leaflets consulted
Headings of leaflets consulted | Month 6
  Headings of leaflets consulted
Number of cards consulted | Month 6
  Number of cards consulted
Headings of cards consulted | Month 6
  Headings of cards consulted
Number of videos consulted | Month 6
  Number of videos consulted
Headings of videos consulted | Month 6
  Headings of videos consulted
Number of address consulted in the address list | Month 6
  Number of address consulted in the address list
Number of upcoming events consulted | Month 6
  Number of upcoming events consulted

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No